CLINICAL TRIAL: NCT05097105
Title: Role of Diffusion -Weighted MRI in Evaluation of Urinary Bladder Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Refaat Abdellah, Assistant lecture of Radiology, Sohag University
Other Study IDs: Soh-Med-21-10-32
Record Dates: First submitted 2021-10-17; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Urinary Bladder Neoplasm
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- urilogic patients
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI sequences: TI. T2 and diffusion weighted

SUMMARY:
Urinary bladder cancer is a common malignant tumor of the urinary tract in both men and women. Proper management of the urinary bladder cancer depends on the stage of the lesions.

Differentiating the histopathological types, tumor grade and the depth of tumor invasion are very important for determining the therapeutic approach and are highly correlated with the recurrence, progression and patient's survival.

Radical cystectomy (RC) and lymphadenectomy after neoadjuvant chemotherapy is the standard treatment for muscle invasive tumors, whereas the treatment of choice for non-muscle invasive tumors is transurethral resection (TUR) ±chemo/immunotherapy.

Cystoscopy with biopsy is still the best tool for bladder cancer staging due to its high sensitivity in detecting lesions and the possibilities of tumor resections, but the main drawbacks are invasiveness, limitation in detection of flat lesions, and lack of the assessment of extra-vesical tumor invasion. Modern diagnostic modalities circumvent these limitations like blue-light cystoscopic examination and infrared cystoscopy.

For the radiological evaluation of the urinary bladder, magnetic resonance imaging (MRI) is a valuable imaging modality due to high tissue contrast and multiplanar imaging capabilities.

Diffusion-weighted images provides useful information for evaluation of local T stage of the urinary bladder cancer, specially in differentiating T1 stage or lower tumors from T2 stage and higher tumor stages.

Apparent diffusion coefficient (ADC) delineating the degree of water molecular diffusion and the degree of restriction to water diffusion in biological tissues is inversely correlated to the integrity of the cell membranes and the tissue cellularity.

The apparent diffusion coefficient (ADC) value has been revealed as quantitative measure of the degree of malignancy of the lesions. Decreased ADC values were reported with malignant lesions which have a larger cell diameter and more cellularity than normal tissue.

ELIGIBILITY:
Inclusion Criteria :• Age, any age will be included

* Sex, both genders are included.
* Patient presenting with heamaturia or intractable cystitis and urinary bladder mass lesions detected on ultrasound and/or CT examinations (with contrast).

Exclusion Criteria:

• General contraindications to MR imaging (pacemaker, metallic prostheses and clostrophobia).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient presenting with heamaturia or intractable cystitis and urinary bladder mass lesions detected on ultrasound and/or CT examinations (with contrast).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of urinary bladder masses | 2 years
  detection and grading of urinary bladder masses using ADC value and pattern of signal of restriction in diffusion weighted image .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Daneshmand S, Bazargani ST, Bivalacqua TJ, Holzbeierlein JM, Willard B, Taylor JM, Liao JC, Pohar K, Tierney J, Konety B; Blue Light Cystoscopy with Cysview Registry Group. Blue light cystoscopy for the diagnosis of bladder cancer: Results from the US prospective multicenter registry. Urol Oncol. 2018 Aug;36(8):361.e1-361.e6. doi: 10.1016/j.urolonc.2018.04.013. Epub 2018 May 30. PMID 29859728
- [Background] Koh DM, Collins DJ. Diffusion-weighted MRI in the body: applications and challenges in oncology. AJR Am J Roentgenol. 2007 Jun;188(6):1622-35. doi: 10.2214/AJR.06.1403. PMID 17515386
- [Background] Green DA, Rink M, Hansen J, Cha EK, Robinson B, Tian Z, Chun FK, Tagawa S, Karakiewicz PI, Fisch M, Scherr DS, Shariat SF. Accurate preoperative prediction of non-organ-confined bladder urothelial carcinoma at cystectomy. BJU Int. 2013 Mar;111(3):404-11. doi: 10.1111/j.1464-410X.2012.11370.x. Epub 2012 Jul 13. PMID 22805163
- [Background] Amin MF, Abd El Hamid AM. The diagnostic accuracy of multidetector computed tomography with multiplanar reformatted imaging and virtual cystoscopy in the early detection and evaluation of bladder carcinoma: comparison with conventional cystoscopy. Abdom Imaging. 2013 Feb;38(1):184-92. doi: 10.1007/s00261-012-9902-6. PMID 22623028